

#### Protocol C3421038

# A PHASE 1, OPEN-LABEL STUDY TO EVALUATE THE PHARMACOKINETIC INTERACTIONS BETWEEN PF-06882961 AND PF-06865571 IN HEALTHY ADULT PARTICIPANTS (PART A) AND OVERWEIGHT ADULTS OR ADULTS WITH OBESITY WHO ARE OTHERWISE HEALTHY (PART B)

Statistical Analysis Plan (SAP)

Version: 2

**Date:** 07-Jul-2021



### TABLE OF CONTENTS

| LIST OF TABLES | 4 |
|------------------------------------------------------------------|----|
| LIST OF FIGURES | |
| APPENDICES | 5 |
| 1. VERSION HISTORY | 6 |
| 2. INTRODUCTION | 6 |
| 2.1. Study Objectives, Endpoints, and Estimands | 7 |
| 2.1.1. Primary Estimand(s) | 8 |
| 2.1.2. Secondary Estimand(s) | 8 |
| 2.1.3. Additional Estimand(s) | 8 |
| 2.2. Study Design | 8 |
| 2.2.1. Treatment Scheme for Part A | 9 |
| 2.2.2. Treatment Scheme for Part B | 9 |
| 3. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS | 10 |
| 3.1. Primary Endpoint(s) | 10 |
| 3.2. Secondary Endpoint(s) | 11 |
| 3.2.1. Safety Endpoints | 11 |
| 3.2.2. Assessment of Mental Health (Part B Only) | 12 |
| 3.2.2.1. Columbia Suicide Severity Rating Scale (C-SSRS) | 12 |
| 3.2.2.2. Patient Health Questionnaire (PHQ-9) | 12 |
| 3.2.3. Other Safety Endpoints (Part B only) | |
| 3.3. Tertiary Endpoint(s) | |
| 3.4. Baseline Variables | 13 |
| 4. ANALYSIS SETS (POPULATIONS FOR ANALYSIS) | 13 |
| 5. GENERAL METHODOLOGY AND CONVENTIONS | 15 |
| 5.1. Hypotheses and Decision Rules | 15 |
| 5.2. General Methods | |
| 5.2.1. Analyses for Binary Endpoints | 15 |
| 5.2.2. Analyses for Continuous Endpoints | 15 |



| 5.2.3. Analyses for Categorical Endpoints | 15 |
|---|---|
| 5.3. Methods to Manage Missing Data | 15 |
| 5.3.1. Pharmacokinetic Concentrations Below the Limit of Quantification | 15 |
| 5.3.2. Deviations, Missing Concentrations and Anomalous Values | 15 |
| 5.3.3. Pharmacokinetic Parameters | 16 |
| 5.3.4. 4-β-hydroxycholesterol, cholesterol and Coproporphyrins I Concentrations and Parameters | 16 |
| 6. ANALYSES AND SUMMARIES | 16 |
| 6.1. Primary Endpoint | 16 |
| 6.1.1. PF-06882961 PK Parameters | 16 |
| 6.1.1.1. Effects of PF-06865571 on Single Dose PF-06882961 PK<br>Parameters (Part A) | 18 |
| 6.1.1.2. Effect of PF-06865571 on the Multi-Dose of PF-06882961 PK Parameters (Part B) | 19 |
| 6.1.2. PF-06865571 PK Parameters | 19 |
| 6.1.2.1. Effect of PF-06882961 on Single Dose PF-06865571 PK Parameters (Part B) | 21 |
| CCI | |
| 6.2. Secondary Endpoint(s) | 21 |
| 6.2.1. Demographic and Physical Examination Data | 21 |
| 6.2.2. Discontinuation(s) | 22 |
| 6.2.3. Adverse Events | 22 |
| 6.2.4. Hypoglycemia (Part B only) | 22 |
| 6.2.5. Laboratory Data | 22 |
| 6.2.6. Vital Signs Data | 22 |
| 6.2.7. Electrocardiogram (ECG) | 23 |
| 6.2.8. C-SSRS (Part B Only) | 23 |
| 6.2.9. PHQ-9 (Part B only) | 23 |
| 6.3. Other Endpoint(s) | 24 |
| 6.3.1. Change from Baseline in PT, INR, aPTT (Part B only) | 24 |



| 6.3 | 3.2. Change from Baseline in TSH, Lipids (Part B only) | 24 |
|---|---|---|
| 6.3 | 3.3. Change from Baseline in Free T4, Calcitonin, Amylase, Lipase, TBA (Part B only) | |
| 6.3 | 3.4. Change from Baseline in Body Weight (Part B Only) | 24 |
| 6.3 | 3.5. Coproporphyrins I (Part B) | 24 |
| 6.3 | 3.6. 4-β-hydroxycholesterol/Cholesterol Ratio | 26 |
| 6.4. Sub | set Analyses | 27 |
| 6.5. Base | eline and Other Summaries and Analyses | 27 |
| 6.5 | 5.1. Baseline Summaries | 27 |
| 6.5 | 5.2. Study Treatment Exposure | 27 |
| C | CI | |
| 6.5 | 5.4. Screening and Other Special Purpose Data | 27 |
| 7. INTERIM A | ANALYSES | 27 |
| 8. REFERENCE | CES | 27 |
| 9. APPENDIC | ES | 28 |
| | LIST OF TABLES | |
| Table 1. | Summary of Changes | 6 |
| Table 2. | Part A – Plasma PK Parameters for PF-06882961 | 10 |
| Table 3. | Part B – Plasma PK Parameters for PF-06882961 CCl and PF-06865571 | 10 |
| Table 4. | Part B – Plasma CP-I Parameters | 13 |
| Table 5. | PF-06882961 and CCl PK Parameters to be Summarized Descriptively per Day. | 17 |
| Table 6. | PF-06865571 PK Parameters to be Summarized Descriptively | 19 |
| Table 7. | CP-I Parameters to be Summarized Descriptively per Day | 25 |

### LIST OF FIGURES

No table of figures entries found.



# **APPENDICES**

| Appendix 1. Summary of Efficacy Analyses | 29 |
|---|---|
| Appendix 2. Data Derivation Details | 29 |
| Appendix 2.1. Definition and Use of Visit Windows in Reporting | 29 |
| Appendix 2.2. Endpoint Derivations | 29 |
| Appendix 2.3. Example SAS Code for Statistical Analyses | 29 |
| Appendix 2.3.1. Analysis for DDI interaction (Part A): | 29 |
| Appendix 2.3.2. Analysis for DDI interaction (Part B): | 29 |
| Appendix 3. List of Abbreviations | 30 |
| Appendix 4. Categorical Classes for ECG and Vital Signs of Potential Clinical Concern | 34 |
| Appendix 5. C-SSRS Mapped to C-CASA - Suicidal Ideation and Behavior Events and Codes | 35 |



#### 1. VERSION HISTORY

**Table 1. Summary of Changes** 

| Version/<br>Date | Associated Protocol / Amendment | Rationale | Specific Changes |
|---|---|---|---|
| 1<br>07-Apr-2021 | Protocol Amendment 1<br>12-Mar-2021 | N/A | N/A |
| 2<br>07-Jul-2021 | Protocol Amendment 2<br>03-Jun-2021 | Preliminary draft data from study C3421007 indicate that a decrease in exposure of midazolam are observed when co-administered with PF-06882961. To investigate the mechanism of this interaction, assessment of plasma 4-β-hydroxycholesterol/cho lesterol, an endogenous probe for CYP3A induction, is being added in Part B. In vitro studies indicate PF-06882961 may inhibit OATP1B1 at dose(s) evaluated in this study. Therefore, to evaluate this potential effect of PF-06882961, measurement of plasma CP-I, an endogenous probe for OATP1B activity, is being added in Part B. | Section 2.1 modified to introduce endogeneous endpoints, Sections 3.3, 5.3.4, 6.3.5 and 6.3.6 created to specify the analyses and reporting of the endogeneous endpoints. Appendix 4 modified to introduce acronyms related to the enedgoneous endpoints |

#### 2. INTRODUCTION

This study will evaluate the PK interactions between PF-06882961 and PF-06865571 in healthy adult participants (Part A) and overweight adults or adults with obesity who are otherwise healthy (Part B).



This statistical analysis plan (SAP) provides the *detailed methodology for summary and* statistical analyses of the data collected in Study C3421038. This document may modify the plans outlined in the protocol; however, any major modifications of the primary endpoint definition or its analysis will also be reflected in a protocol amendment.

#### 2.1. Study Objectives, Endpoints, and Estimands

| Objectives | Endpoints |
|---|---|
| Part A | |
| Primary: | Primary: |
| To evaluate the effects of PF-06865571 on the single-dose pharmacokinetics of PF-06882961 in healthy adult participants. | PF-06882961 plasma pharmacokinetic parameters: C <sub>max</sub> and AUC <sub>24</sub> . |
| Secondary: | Secondary: |
| To evaluate the safety and tolerability of PF-06882961 alone and in combination with PF-06886571 when administered to healthy adult participants. | Assessment of treatment-emergent adverse events, clinical laboratory abnormalities, vital signs, body weight, and ECG parameters during the entire study. |
| Tertiary/Exploratory: | Tertiary/Exploratory: |
| To evaluate the effects of PF-06865571 on additional pharmacokinetic parameters of PF-06882961 in healthy adult participants. | Additional PF-06882961 plasma pharmacokinetic parameters: $T_{max}$ . |
| Part B | |
| Primary: | Primary: |
| To evaluate the effects of PF-06882961 on the single-dose pharmacokinetics of PF-06865571 in overweight adults or adults with obesity who are otherwise healthy. | PF-06865571 plasma pharmacokinetic parameters on Day 1 and Day 47: $C_{max}$ , $AUC_{last}$ , and $AUC_{inf}$ , as data permits. |
| To evaluate the effects of PF-06865571 on the multiple-dose pharmacokinetics of PF-06882961 in overweight adults or adults with obesity who are otherwise healthy. | PF-06882961 plasma pharmacokinetic parameters on Day 46 and Day 61: $C_{max}$ and $AUC_{12}$ . |
| Secondary: | Secondary: |
| To evaluate the safety and tolerability of PF-06882961 and PF-06865571 when administered separately and in combination in overweight adults or adults with obesity who are otherwise healthy. | Assessment of treatment-emergent adverse events, clinical laboratory abnormalities, vital signs, body weight, and ECG parameters during the entire study. |
| | Assessment of mental health as determined by C-SSRS and PHQ-9 in Part B of this study. |
| To evaluate the effects of PF-06882961 on | Tertiary/Exploratory: Additional PF-06865571 plasma pharmacokinetic |
| additional pharmacokinetic parameters of PF-06865571 in overweight adults or adults with obesity who are otherwise healthy. | parameters on Day 1 and Day 47: $T_{max}$ , CL/F, $V_z/F$ , and $t_{1/2}$ , as data permits. |



To evaluate the effects of PF-06865571 on additional pharmacokinetic parameters of PF-06882961 in overweight adults or adults with obesity who are otherwise healthy.

Additional PF-06882961 plasma pharmacokinetic parameters on Day 46 and Day 61: T<sub>max</sub> and CL/F.



To evaluate the effects of PF-06882961 on the multiple-dose pharmacokinetics of PF-06865571 in overweight adults or adults with obesity who are otherwise healthy.

To evaluate the effects of multiple doses of PF-06882961 on CYP3A induction in overweight adults or adults with obesity who are otherwise healthy.

To evaluate the effect of multiple doses of PF-06882961 on coproporphyrins I in overweight adults or adults with obesity who are otherwise healthy.

PF-06865571 plasma pharmacokinetic parameters on Day 61:  $C_{max}$ ,  $T_{max}$ , and  $AUC_{12}$ .

Morning pre-dose 4- $\beta$ -hydroxycholesterol/cholesterol plasma ratio on Days 1, 19, 31, and 47.

CP-I parameters on Days 30 and 46: AUC<sub>12</sub> and C<sub>max</sub>.

#### 2.1.1. Primary Estimand(s)

Not applicable

#### 2.1.2. Secondary Estimand(s)

Not applicable

#### 2.1.3. Additional Estimand(s)

Not applicable

#### 2.2. Study Design

*This study will be conducted in 2 parts.* 

**Part A** is an open-label, two-period, two-sequence, crossover cohort investigating the potential effect of PF-06865571 on the PK of PF-06882961 in healthy adult participants. **Part B** is an open-label, fixed-sequence cohort to evaluating the effect of PF-06882961 on the PK of PF-06865571, as well as the effect of PF-06865571 on the PK of PF-06882961 in overweight adults or adults with obesity who are otherwise healthy. The effect of PF-06882961 on PF-06865571 PK will be evaluated at steady-state at a dose of up to 200 mg BID of PF-06882961. Then, PF-06882961 and PF-06865571 will be coadministered for approximately 2 weeks for further evaluation of PK interactions and to generate additional safety and tolerability data on the combination.



A cohort of approximately 8 participants will be enrolled in Part A. Approximately 16 participants will be enrolled in Part B such that approximately 12 evaluable participants complete Part B.

#### 2.2.1. Treatment Scheme for Part A

| | Period 1 | Washout* | Period 2 |
|---|---|---|---|
| Sequence 1 (n=4) | Treatment A:<br>20 mg PF-06882961 single dose | Washout of at<br>least 3 days* | Treatment B:<br>20 mg PF-06882961 single dose<br>plus<br>300 mg PF-06865571 single dose |
| Sequence 2 (n=4) | Treatment B:<br>20 mg PF-06882961 single dose<br>plus<br>300 mg PF-06865571 single dose | Washout of at<br>least 3 days* | Treatment A:<br>20 mg PF-06882961 single dose |

<sup>\*</sup>Each participant is planned to undergo 2 treatment periods with a washout interval between periods of at least 3 days following the final dose of study intervention administered in Period 1.

#### 2.2.2. Treatment Scheme for Part B

| | Period 1 | Period 2 | Period 3 | Period 4 |
|---|---|---|---|---|
| | Days 1-2 | Days 3-46 | Days 47-48 | Days 49-62 |
| PF-06865571<br>(DGAT2)<br>Dose | 300 mg single dose<br>on Day 1 only <sup>a</sup> | N/A | 300 mg single dose<br>on Day 47 only <sup>a</sup> | 300 mg BID<br>on Days 49-61 <sup>a</sup> |
| PF-06882961<br>(GLP-1)<br>Dose | N/A | 10 mg BID titrated to 200 mg BID <sup>b,c</sup> | 200 mg BID <sup>c</sup> | 200 mg BID<br>on Days 49-61 <sup>b,c</sup> |

a. Dense PK sampling for measurement of PF-06865571 plasma concentrations on Day 1 (reference), Day 47 (test), and Day 61 (summary statistics only).

In all study parts (Part A and Part B), participants will remain on-site (inpatient study) for the duration of the dosing period, followed by one follow-up outpatient visit. A further follow-up contact with participants will be conducted at least 28 days and up to 35 days after the last administration of IP; this contact may be done via a phone call.

The study will be conducted in the US.

b. Dense PK sampling for measurement of PF-06882961 plasma concentrations on Day 46 (reference) and Day 61 (test).

c. Doses of PF-06882961 may be reduced based on PK results of Part A of this study and safety and tolerability results of Study C3421007.



Participants who discontinue prior to completion of the study may be replaced, at the discretion of the principal investigator (PI) and sponsor (applicable to part A only).

# 3. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS

#### 3.1. Primary Endpoint(s)

Blood samples for PK analysis of PF-06865571, PF-06882961 CCl will be taken according to the Schedule of Activities (SoA) given in the protocol.

In Part A, plasma PF-06882961 PK parameters following single administration of PF-06882961 will be derived using standard noncompartmental methods, as data permit, for each treatment, from the concentration time profiles as follows:

Table 2. Part A – Plasma PK Parameters for PF-06882961

| Parameter | Analysis Scale | PF-06882961 |
|-------------------|----------------|-------------|
| AUC <sub>24</sub> | ln | D |
| $C_{max}$ | ln | D |
| $T_{max}$ | R | D |

Key: D=displayed with descriptive statistics, ln=natural-log transformed, R=raw (untransformed)

In Part B, plasma PF-06865571, PF-06882961, PK parameters following single administration of PF-06865571 and PF-06882961 or multiple-dose of PF-06882961 will be derived using standard noncompartmental methods, as data permit, for each treatment and day (as appropriate), from the concentration time profiles as follows:

Table 3. Part B – Plasma PK Parameters for PF-06882961, CCl and PF-06865571

| Parameter | Compound CCI | Days | Analysis<br>Scale | Reporting |
|---|---|---|---|---|
| AUClast | PF-06865571 | 1 and 47 | ln | D |
| AUCinf* | PF-06865571 | 1 and 47 | ln | D |
| AUC <sub>12</sub> | PF-06865571 | 61 | ln | D |
| | PF-06882961 CCI | 46 and 61 | | |
| Cmax | PF-06865571 | 1, 47, and 61 | ln | D |
| | PF-06882961 CCI | 46 and 61 | | |
| Tmax | PF-06865571 | 1, 47, and 61 | R | D |
| | PF-06882961 CCI | 46 and 61 | | |



| t1/2* | PF-06865571 | 1 and 47 | R | D |
|-------|-------------|-----------|----|---|
| CL/F* | PF-06865571 | 1 and 47 | ln | D |
| | PF-06882961 | 46 and 61 | | |
| Vz/F* | PF-06865571 | 1 and 47 | ln | D |

#### CCI

Key: D=displayed with descriptive statistics, ln=natural-log transformed, R=raw (untransformed), \*=if data permits

#### 3.2. Secondary Endpoint(s)

#### 3.2.1. Safety Endpoints

• Assessment of treatment-emergent adverse events, clinical laboratory abnormalities, vital signs, body weight and ECG parameters during the entire study.

Any events occurring following start of study intervention (i.e. treatment) will be counted as treatment emergent.

Events that occur in a non-treatment period (for example, Washout or Follow-up) will be counted as treatment emergent and attributed to the most recent treatment taken.

A 3-tier approach for summarizing adverse events (AEs) will not be used due to the low number of participants planned to be recruited.

The following data are considered in standard safety summaries (see protocol for collection days and list of parameters):

- adverse events,
- laboratory data,
- vital signs data,
- body weight
- ECG results.

For laboratory, vital signs and ECG data there will be two separate definitions for baseline that will be calculated depending on the study part:

- i) For Part A, using the last pre-dose measurement within each respective treatment Period
- ii) For Part B, using a fixed baseline of the last pre-dose measurement in Period 1.



Change from baseline will therefore be calculated twice for each relevant safety endpoint using (i) and (ii) above.

Definitions of baseline body weight for exploratory safety analyses are described in Section 3.2.3.

#### 3.2.2. Assessment of Mental Health (Part B Only)

• Assessment of mental health as determined by C-SSRS and PHQ-9 during the entire study.

#### 3.2.2.1. Columbia Suicide Severity Rating Scale (C-SSRS)

The C-SSRS is a validated tool to evaluate suicidal ideation and behavior. Data relevant to the assessment of suicidality will be mapped to the Columbia-Classification Algorithm of Suicide Assessment (C-CASA) codes as given in Appendix 5.

Baseline is defined as the last pre-dose measurement in Period 1. For this endpoint the screening visit will be labelled as 'Lifetime' in tables and the recent history (i.e. past 12 months) will also be reported separately.

#### 3.2.2.2. Patient Health Questionnaire (PHQ-9)

The PHQ-9 is a 9 item self-report scale for the assessment of depressive symptoms. The PHQ-9 will be completed by participants and reviewed by site staff at the pre-defined time points outlined in the SoA for Part B.

Baseline is defined as the last pre-dose measurement in Period 1 Day 1.

#### 3.2.3. Other Safety Endpoints (Part B only)

• Change from baseline in PT/INR/aPTT, TBA, HbA1c, body weight, lipids, TSH, Free T4, calcitonin, amylase, and lipase at all post-dose time points as outlined in the SoA for Part B.

Baseline is defined as the last pre-dose measurement in Period 1 Day 1.

#### 3.3. Tertiary Endpoint(s)

In Part B, plasma samples for analysis of  $4-\beta$ -hydroxycholesterol/cholesterol ratio and CP-I concentrations will be taken according to the Schedule of A.

Plasma CP-I parameters will be derived using standard noncompartmental methods, as data permit, for each treatment and day (as appropriate), from the concentration time profiles as follows:



| Table 4. | Part R _ | Plasma | CP-I | <b>Parameters</b> |
|----------|--------------|-------------|--------|-------------------|
| I am T. | 1 41 1 1 7 - | ' i iasilia | V 1 -1 | i ai aiiicteis |

| Parameter | Marker | Days | Analysis<br>Scale | Reporting |
|---|---|---|---|---|
| AUC <sub>12</sub> | CP-I | 30 and 46 | ln | D |
| Cmax | CP-I | 30 and 46 | ln | D |
| Key: D=displayed with descriptive statistics, ln=natural-log transformed | | | | |

#### 3.4. Baseline Variables

Baseline for all parameters discussed in Section 5 and 6 will be defined as the values assessed on as the closest measurement before dosing (ie pre-dose on Day 1 0H).

When three assessements are performed at baseline, the baseline will be the average of the three values (eg Vital Signs).

#### 4. ANALYSIS SETS (POPULATIONS FOR ANALYSIS)

Data for all participants will be assessed to determine if participants meet the criteria for inclusion in each analysis population prior to releasing the database and classifications will be documented per standard operating procedures.

All analyses will be performed on an "as-treated" basis and will not include data from participants who are randomized but not treated. If a participant takes a treatment that is not consistent with the treatment they are randomized to, for example takes a treatment out of sequence or takes the same treatment twice, then they will be reported under the treatment that they actually receive for all safety, PK and PD analyses, where applicable.

Participants who experience events that may affect their PK profile (eg vomiting) may be excluded from the PK analysis. At the discretion of the pharmacokineticist a concentration value may also be excluded if the deviation in sampling time is of sufficient concern or if the concentration is anomalous for any other reason.

A full list of protocol deviations (eg medication errors) will be compiled and reviewed to identify major and minor deviations prior to database closure.

| Population | Description |
|---|---|
| Enrolled | All participants who sign the ICD. |
| Randomly assigned to investigational product | All participants randomly assigned to investigational product regardless of whether or not the investigational product was administered. |



| Population | Description |
|---|---|
| Evaluable | All participants randomly assigned to investigational product and who take at least 1 dose of investigational product. Participants will be analyzed according to the product they actually received. |
| Safety | All participants randomly assigned to investigational product and who take at least 1 dose of investigational product. Participants will be analyzed according to the product they actually received. |
| PF-06865571 PK<br>Concentration Set | The PF-06865571 PK concentration population is defined as all randomized participants who received at least 1 dose of PF-06865571 and in whom at least 1 plasma concentration value is reported. |
| PF-06865571 PK<br>Parameter Set | The PF-06865571 PK parameter population is defined as all randomized participants who received at least 1 dose of PF-06865571 and in whom at least 1 parameter value is reported. |
| PF-06882961<br>PK Concentration Set | The PF-06882961 concentration population is defined as all randomized participants who received at least 1 dose of PF-06882961 and in whom at least 1 plasma concentration value is reported. |
| PF-06882961<br>PK Parameter Set | The PF-06882961 PK parameter population is defined as all randomized participants who received at least 1 dose of PF-06882961 and in whom at least 1 parameter value is reported. |
| Endogenous biomarker<br>Concentration Set | The endogenous biomarker concentration population is defined as all randomized participants who received at least 1 dose of PF-06882961 and in whom at least 1 plasma concentration (4-β-hydroxycholesterol and cholesterol or CP-I) value is reported. |
| Endogenous biomarker<br>Parameter Set | The endogenous biomarker parameter population is defined as all randomized participants who received at least 1 dose of PF-06882961 and in whom at least 1 CP-I or 4-β-hydroxycholesterol/cholesterol parameter value is reported. |



#### 5. GENERAL METHODOLOGY AND CONVENTIONS

#### 5.1. Hypotheses and Decision Rules

Not applicable

#### **5.2.** General Methods

#### 5.2.1. Analyses for Binary Endpoints

Not applicable

#### **5.2.2.** Analyses for Continuous Endpoints

Continuous endpoints and relevant safety endpoints will be presented using summary statistics: number of observations, arithmetic mean, standard deviation, median, minimum and maximum values.

#### 5.2.3. Analyses for Categorical Endpoints

Categorical endpoints and relevant safety endpoints will be presented using summary statistics: number of observations, counts and percentages.

#### 5.3. Methods to Manage Missing Data

For the analysis of safety endpoints, the sponsor data standard rules for imputation will be applied.

In all exploratory safety data presentations (except listings), concentrations below the limit of quantification (BLQ) will be set to the lower limit of quantification (LLQ).

#### 5.3.1. Pharmacokinetic Concentrations Below the Limit of Quantification

In all PK data presentations (except listings), concentrations below the limit of quantification (BLQ) will be set to zero. In listings BLQ values will be reported as "<LLOQ", where LLOQ will be replaced with the value for the lower limit of quantification.

#### 5.3.2. Deviations, Missing Concentrations and Anomalous Values

In PK summary tables and plots of median profiles, statistics will be calculated having set concentrations to missing if 1 of the following cases is true:

- 1. A concentration has been collected as ND (ie, not done) or NS (ie, no sample),
- 2. A deviation in sampling time is of sufficient concern or a concentration has been flagged anomalous by the pharmacokineticist/clinical team.

Note that summary statistics will not be presented at a particular time point if more than 50% of the data are missing.



Participants who experience events that may affect their PK profile (e.g. lack of compliance with dosing or vomiting) may be excluded from the PK analysis. At the discretion of the pharmacokineticist a concentration value may also be excluded if the deviation in sampling time is of sufficient concern or if the concentration is anomalous for any other reason.

A full list of protocol deviations will be compiled and reviewed to identify major and minor deviations prior to database closure.

#### 5.3.3. Pharmacokinetic Parameters

Actual PK sampling times will be used in the derivation of PK parameters.

If a PK parameter cannot be derived from a participant's concentration data, the parameter will be coded as NC (ie, not calculated). Note that NC values will not be generated beyond the day that a participant discontinues.

In summary tables, statistics will be calculated by setting NC values to missing; and statistics will be presented for a particular dose with  $\geq 3$  evaluable measurements.

If a participant receives a dose that was not assigned based on the randomized titration scheme (for example due to a down-titration), the PK data from that Day will not be included in the calculation of summary statistics but will be included in listings.

If an individual participant has a known biased estimate of a PK parameter (due for example to an unexpected event such as vomiting before all the compound is adequately absorbed in the body), this will be footnoted in summary tables and will not be included in the calculation of summary statistics or statistical analyses.

# 5.3.4. 4-β-hydroxycholesterol, cholesterol and Coproporphyrins I Concentrations and Parameters

Rules described in Section 5.3.1, and Section 5.3.2 will be used to manage concentrations below limit of quantification, deviations, missing concentrations and anomalous value for the markers of CYP3-A induction (ie 4-β-hydroxycholesterol/cholesterol ratio), and OATP1B1 Activity (ie coproporphyrins I).

Rules described in Section 5.3.3 will apply to derive parameters for Coproporphyrins I (CP-I) and 4-β-hydroxycholesterol/cholesterol ratio.

#### 6. ANALYSES AND SUMMARIES

#### 6.1. Primary Endpoint

#### 6.1.1. PF-06882961 PK Parameters

Applicable to Parts A, and B – Analyses reported for each part separately.



- Estimand strategy: Not applicable
- Analysis set: PF-06882961 Concentration and Pharmacokinetic Parameter Set

To assess the pharmacokinetics of PF-06882961 in Part A and Part B CCI the PK parameters detailed in Section 3.1 will be listed and summarized for participants in the PK analysis set (as defined in Section 4). Missing values will be handled as detailed in Section 5.3 along with handling of values where participants received a dose that was not assigned based on the titration scheme). Each PK parameter will be summarized by treatment (eg differentiating different doses and dosing frequencies as required), Study Part and Study Day/Period (as appropriate).

The parameters will include the set of summary statistics as specified in the table below:

Table 5. PF-06882961 CC PK Parameters to be Summarized Descriptively per Day

| Part | Parameter | Days | Summary Statistics |
|---|---|---|---|
| A | AUC <sub>24</sub> , C <sub>max</sub> | - | N, arithmetic mean, median, cv%, standard |
| | | | deviation, minimum, maximum, geometric |
| | | | mean and geometric cv%. |
| | T <sub>max</sub> | - | N, median, minimum, maximum. |
| В | $AUC_{12}, C_{max},$ | 46 and 61 | N, arithmetic mean, median, cv%, standard |
| | CCI CL/F* | | deviation, minimum, maximum, geometric |
| | | | mean and geometric cv%. |
| | T <sub>max</sub> | 46 and 61 | N, median, minimum, maximum. |

\* if data permits

There will be one summary table presenting all PK parameters. The treatment subheading will include the study part, analyte, dose information and day (Day 46 or Day 61). As per Section 5.3.3, data collected on days that participants received anything other than the assigned dose based on the titration scheme will only be listed and not summarized as part of the summary table.

The following plots will be presented:

- Box and whisker plots for individual PK parameters of PF-06882961 (AUC<sub>24</sub>, and C<sub>max</sub>) will be presented by treatment and overlaid with geometric means for Part A.
- Box and whisker plots for individual PK parameters of PF-06882961 (AUC<sub>12</sub>, C<sub>max</sub>) will be presented by treatment and overlaid with geometric means for Part B.

Presentations for PF-06882961 CCl concentrations will include:



- a listing of all concentrations sorted by participant ID, treatment, and matrix and nominal time postdose. The concentration listing will also include the actual times. Deviations from the nominal time will be given in a separate listing.
- a summary of concentrations by treatment, and nominal time postdose, where the set of statistics will include n, mean, median, standard deviation, coefficient of variation (cv), minimum, maximum and the number of concentrations above the lower limit of quantification.
- median concentration time plots (on both linear and semi-log scales) against nominal time post-dose by treatment period. One plot for each scale will be presented which will include the different PF-06882961 treatment periods in the same plot.
- mean concentrations time plots (on both linear and semi-log scales) against nominal time post-dose by treatment period. One plot for each scale will be presented which will include the different PF-06882961 treatment periods in the same plot.
- individual concentration time plots by treatment period (on both linear and semi-log scales) against actual time post-dose (there will be separate spaghetti plots for each treatment period, with a line for each participant per scale).

The length of time used for the x-axes of these plots will be decided on review of the data, and will depend on how long PF-06882961 concentration is quantifiable in the plasma.

For summary statistics, median and mean plots by sampling time, the nominal PK sampling time will be used, for individual participant plots by time, the actual PK sampling time will be used.

#### 6.1.1.1. Effects of PF-06865571 on Single Dose PF-06882961 PK Parameters (Part A)

Natural log-transformed  $C_{max}$  and  $AUC_{24}$  of PF-06882961 administered alone or co-administered with PF-06865571 will be analyzed using a mixed effect model with treatment, sequence, and period as a fixed effects and participant embedded in sequence as a random effect. The Kenward-Roger approximation will be used for estimating degrees of freedom for the model parameters. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals will be obtained from the models. The adjusted mean differences and 90% confidence intervals for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios. The reference treatment will be "PF-06882961 20 mg plus PF-06865571 300 mg BID"



# 6.1.1.2. Effect of PF-06865571 on the Multi-Dose of PF-06882961 PK Parameters (Part B)

To analyze the effects of PF-06865571 on multi-dose PF-06882961 PK parameters, *natural log-transformed AUC*<sub>12</sub> *and C*<sub>max</sub> *of PF-06882961* 200 mg *BID administered alone* (Period 2 – Day 46) *or co-administered with PF-06865571* 300 mg *BID* (Period 4 – Day 61) *will be analyzed* using a mixed effect model including treatment as fixed effects and participant as random effect. The Kenward-Roger approximation will be used for estimating degrees of freedom for the model parameters. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals will be obtained from the models. The adjusted mean differences and 90% confidence intervals for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios. *The test treatment will be* "PF-06865571 300 mg BID plus PF-06882961 200 mg BID" (Period 4 – Day 61), which will be reported separately in comparison to the reference treatment of "PF-06882961 200 mg BID administered alone" (Period 2 – Day 46).

#### 6.1.2. PF-06865571 PK Parameters

Applicable to Part B only.

• Estimand strategy: Not applicable

• Analysis set: PF-06865571 Concentration and Pharmacokinetic Parameter Set

To assess the pharmacokinetics of PF-06865571, the PK parameters detailed in Section 3.1 will be listed and summarized for participants in the PK analysis set (as defined in Section 4). Missing values will be handled as detailed in Section 5.3 along with handling of values where participants received a dose that was not assigned based on the titration scheme). Each PK parameter will be summarized by treatment (eg differentiating different doses and dosing frequencies as required), and Study Day as applicable.

The parameters will include the set of summary statistics as specified in the table below:

Table 6. PF-06865571 PK Parameters to be Summarized Descriptively

| Parameter | Days | <b>Summary Statistics</b> |
|---|---|---|
| AUC <sub>last</sub> , AUC <sub>inf</sub> *,<br>CL/F*, Vz/F* | 1 and 47 | N, arithmetic mean, median, cv%, standard deviation, minimum, maximum, |
| | | geometric mean and geometric cv%. |
| $T_{max}$ | 1, 47 and 61 | N, median, minimum, maximum. |
| t <sub>1/2</sub> * | 1, and 47 | N, arithmetic mean, median, cv%, standard deviation, minimum, maximum. |



| C <sub>max</sub> | 1, 47 and 61 | N, arithmetic mean, median, cv%, standard deviation, minimum, maximum, geometric mean and geometric cv%. |
|---|---|---|
| AUC <sub>12</sub> | 61 | N, arithmetic mean, median, cv%, standard deviation, minimum, maximum, geometric mean and geometric cv%. |

<sup>\*</sup> if data permits

There will be one summary table presenting all PK parameters. The treatment subheading will include the analyte, dose information and day (Day 1, Day 47 or Day 61). As per Section 5.3.3, data collected on days that participants received anything other than the assigned dose based on the titration scheme will only be listed and not summarized as part of the summary table.

The following plots will be presented:

• Box and whisker plots for individual PK parameters of PF-06865571 (AUC<sub>last</sub>, AUC<sub>inf</sub>\*, and C<sub>max</sub>) will be presented by treatment and overlaid with geometric means.

Presentations for PF-06865571 concentrations will include:

- a listing of all concentrations sorted by participant ID, treatment, and matrix and nominal time postdose. The concentration listing will also include the actual times. Deviations from the nominal time will be given in a separate listing.
- a summary of concentrations by treatment, and nominal time postdose, where the set of statistics will include n, mean, median, standard deviation, coefficient of variation (cv), minimum, maximum and the number of concentrations above the lower limit of quantification.
- median concentration time plots (on both linear and semi-log scales) against nominal time post-dose by treatment period. One plot for each scale will be presented which will include the different PF-06865571 treatment periods in the same plot.
- mean concentrations time plots (on both linear and semi-log scales) against nominal time post-dose by treatment period. One plot for each scale will be presented which will include the different PF-06865571 treatment periods in the same plot.
- individual concentration time plots by treatment period (on both linear and semi-log scales) against actual time post-dose (there will be separate spaghetti plots for each treatment period, with a line for each participant per scale).



The length of time used for the x-axes of these plots will be decided on review of the data, and will depend on how long PF-06865571 concentration is quantifiable in the matrix.

For summary statistics, median and mean plots by sampling time, the nominal PK sampling time will be used; for individual participant plots by time, the actual PK sampling time will be used.

#### 6.1.2.1. Effect of PF-06882961 on Single Dose PF-06865571 PK Parameters (Part B)

To analyze the effects of PF-06882961 on single-dose PF-06865571 PK parameters, natural log-transformed  $C_{max}$ ,  $AUC_{last}$ , and  $AUC_{inf}$  (as data permit) of PF-06865571 300 mg BID administered alone or co-administered with PF-06882961 will be analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. The Kenward-Roger approximation will be used for estimating degrees of freedom for the model parameters. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals will be obtained from the models. The adjusted mean differences and 90% confidence intervals for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios. The test treatment will be "PF-06865571 300 mg plus PF-06882961 200 mg BID" (Period 3 – Day 47), which will be reported separately in comparison to the reference treatment of "PF-06865571 300 mg" (Period 1 – Day 1).



#### **6.2. Secondary Endpoint(s)**

#### 6.2.1. Demographic and Physical Examination Data

Applicable to Parts A, and B – Analyses reported for each part separately.

A breakdown of demographic data will be provided for age, gender, race, and ethnicity. The physical measurement (weight, body mass index and height) at baseline will also be summarized. Each will be summarized by treatment and 'All Subjects' in accordance with the sponsor reporting standards.

**For Part B only**, an additional table summarizing the screening data of free T4, TSH, calcitonin, amylase, lipase, lipids, PT/INR/aPTT, TBA and HbA1c will be produced as above.





Finally, data collected at screening that are used for inclusion/exclusion criteria, such as laboratory data (unless noted above) will be reported for randomized participants.

#### **6.2.2. Discontinuation(s)**

Applicable to Parts A and B – Analyses reported for each part separately.

Subject discontinuations, temporary discontinuations or dose reductions due to adverse events will be detailed and summarized by treatment.

Data will be reported in accordance with the sponsor reporting standards.

#### **6.2.3.** Adverse Events

Applicable to Parts A, and B – Analyses reported for each part separately:

Adverse events will be reported in accordance with the sponsor reporting standards.

Incidence and severity of treatment emergent adverse event (TEAE) tables will additionally be produced ('All causality' and 'Treatment related', separately) to summarise the total number of adverse events by preferred term, which will be reported by treatment group and overall in accordance with sponsor reporting standards using the safety analysis set defined in Section Section 4

#### 6.2.4. Hypoglycemia (Part B only)

Any hypoglycemic AEs will be listed in a separate table and summarized categorically by treatment as per Section 5.2.3 using the safety population defined in Section 4

#### 6.2.5. Laboratory Data

Applicable to Parts A, and B – Analyses reported for each part separately:

Laboratory data will be listed and summarized by treatment in accordance with the sponsor reporting standards using the safety population defined in Section 4 Baseline is as defined in Section 3.4.

#### 6.2.6. Vital Signs Data

Applicable to Parts A, and B – Analyses reported for each part separately:

Absolute values and change from baseline in supine systolic and diastolic blood pressure and pulse rate will be summarized by treatment, time post-dose and day, according to sponsor reporting standards. Tables will be paged by parameter. Baseline is as defined in Section 3.4.



Mean changes from baseline for supine systolic and diastolic blood pressure and pulse rate will be plotted against time post-dose and day. On each plot there will be 1 line for each treatment.

Maximum absolute values and changes from baseline for vital signs will be summarized descriptively by treatment using categories as defined in Section 5.2.3. Numbers and percentages of subjects meeting the categorical criteria will also be provided. All planned and unplanned post-dose timepoints will be counted in these categorical summaries. All values meeting the criteria of potential clinical concern will be listed.

#### 6.2.7. Electrocardiogram (ECG)

Applicable to Parts A, and B – Analyses reported for each part separately.

Absolute values and changes from baseline in QT interval, heart rate, QTcF interval, PR interval and QRS interval will be summarized by treatment, time postdose, and day using sponsor reporting standards using the safety population defined in Section 4 Tables will be paged by parameter. Baseline is as defined in Section 3.4.

Mean changes from baseline in ECG parameters will be plotted against day. On each plot there will be 1 line for each treatment. Corresponding individual plots of changes from baseline will also be produced for each treatment.

Numbers and percentages of subjects meeting the categorical criteria will be provided. All planned and unplanned post-dose time-points will be counted in these categorical summaries. All values meeting the criteria of potential clinical concern will be listed.

Listings of subjects with any single post-dose value >500 msec will also be produced for QTcF.

QTcB will be listed only and not summarized.

#### 6.2.8. C-SSRS (Part B Only)

Screening, baseline and post-baseline C-SSRS data (mapped to C-CASA scores as described in Section 3.2.2.1) using the safety population defined in Section 4 will be summarized categorically by treatment and time point as outlined in Section 5.2.3.

#### 6.2.9. PHQ-9 (Part B only)

Baseline and post-baseline PHQ-9 data (responses to each of the 9 items) using the safety population defined in Section 4 will be summarized categorically for each question separtely by treatment and time point as outlined in Section 5.2.3.



#### 6.3. Other Endpoint(s)

#### 6.3.1. Change from Baseline in PT, INR, aPTT (Part B only)

• Estimand strategy: Not applicable

• Analysis set: Safety Population Set

Absolute values and change from baseline will be summarized descriptively by treatment and timepoint as described in Section 5.2.2

#### **6.3.2.** Change from Baseline in TSH, Lipids (Part B only)

• Estimand strategy: Not applicable

• Analysis set: Safety Population Set

Absolute values and change from baseline will be summarized descriptively by treatment and timepoint as described in Section 5.2.2

#### 6.3.3. Change from Baseline in Free T4, Calcitonin, Amylase, Lipase, TBA (Part B only)

• Estimand strategy: Not applicable

• Analysis set: Safety Population Set

Absolute values and change from baseline will be summarized descriptively by treatment and timepoint as described in Section 5.2.2

#### 6.3.4. Change from Baseline in Body Weight (Part B Only)

The change from baseline and percent change from baseline to all post-dose timepoints as specified in the SoA will be calculated.

• Estimand strategy: Not applicable

Analysis set: Safety Population Set

Absolute values, change from baseline, and percent change from baseline will be summarized descriptively by treatment and day as per Section 5.2.2

#### 6.3.5. Coproporphyrins I (Part B)

Estimand strategy: Not applicable

Analysis set: Endogenous biomarker Concentration and Parameter Population Set



To assess the effects of PF-06882961 on coproporphyrins I (CP-I) in Part B, the CP-I parameters detailed in Section 3.3 will be listed and summarized for participants in the endogenous biomarker analysis set (as defined in Section 4). Missing values will be handled as detailed in Section 5.3 along with handling of values where participants received a dose that was not assigned based on the titration scheme). Each CP-I parameter will be summarized by treatment (eg differentiating different doses and dosing frequencies as required), Study Part and Study Day/Period (as appropriate).

The parameters will include the set of summary statistics as specified in the table below:

PartParameterDaysSummary StatisticsAUC12, AUC12/12<br/>(ie Cav), Cmax30 and 46N, arithmetic mean, median, cv%, standard deviation, minimum, maximum, geometric mean and geometric cv%.

Table 7. CP-I Parameters to be Summarized Descriptively per Day

On Day 1, individual  $C_{av}$  and individual  $C_{max}$  will be the mean of CP-I plasma concentrations and will serve as baseline to calculate individual change from baseline for each parameter on Day 30 and Day 46. These individual calculated means will also be used for Day1 graphical presentations.

Change from baseline in  $C_{av}$  and  $C_{max}$  for CP-I will be analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect.

Estimates of the adjusted mean differences against the reference will be obtained and corresponding 90% CIs will be reported from the models. The test treatments will be "PF-06882961 120 mg BID" (Day 30) and "PF-06882961 200 mg BID" (Day 46) and reference treatment is "No PF-06882961" (Day 1).

There will be one summary table presenting all parameters. The treatment subheading will include the dose information and day (Day 1, Day 30 or Day 46). As per Section 5.3, data collected on days that participants received anything other than the assigned dose based on the titration scheme will only be listed and not summarized as part of the summary table.

The following plots will be presented:

• Box and whisker plots for individual parameters of CP-I (ie C<sub>av</sub> and C<sub>max</sub>) will be presented by treatment and overlaid with geometric means.

Presentations for CP-I concentrations will include:



- a listing of all concentrations sorted by participant ID, treatment, and nominal time postdose. The concentration listing will also include the actual times. Deviations from the nominal time will be given in a separate listing.
- a summary of concentrations by treatment, and nominal time postdose, where the set of statistics will include n, mean, median, standard deviation, coefficient of variation (cv), minimum, maximum and the number of concentrations above the lower limit of quantification.
- median concentration time plots (on both linear and semi-log scales) against nominal time post-dose by treatment period. One plot for each scale will be presented which will include the different PF-06882961 treatment periods in the same plot.
- mean concentrations time plots (on both linear and semi-log scales) against nominal time post-dose by treatment period. One plot for each scale will be presented which will include the different PF-06882961 treatment periods in the same plot.
- individual concentration time plots by treatment period (on both linear and semi-log scales) against actual time post-dose (there will be separate spaghetti plots for each treatment period, with a line for each participant per scale).

For summary statistics, median and mean plots by sampling time, the nominal blood sampling time will be used; for individual participant plots by time, the actual blood sampling time will be used.

#### 6.3.6. 4-β-hydroxycholesterol/Cholesterol Ratio

The percent change from baseline to all post-dose timepoints as specified in the SoA will be calculated.

- Estimand strategy: Not applicable
- Analysis set: Endogenous biomarker Concentration and Parameter Population Set

Absolute values, and percent change from baseline will be summarized descriptively by treatment and day as per Section 5.2.2

The following plot will be presented:

• Box and whisker plots will be presented by treatment and overlaid with geometric means.



#### 6.4. Subset Analyses

Not applicable.

#### 6.5. Baseline and Other Summaries and Analyses

#### 6.5.1. Baseline Summaries

For each part of the study, and for each endpoint defined in this statistical analysis, baseline assessment will be summarized by treatment as per Section 5.2.2 and Section 5.2.3.

#### **6.5.2. Study Treatment Exposure**

For each part of the study, participant treatment exposure groups will be reported. Frequency counts will be supplied for participant discontinuation(s) by treatment.

Data will be reported in accordance with the sponsor reporting standards.



#### 6.5.4. Screening and Other Special Purpose Data

For each part of the study, prior medication(s) and non-drug treatment(s), serum FSH concentrations, urine drug screen, will be obtained at Screening.

These data will be listed.

#### 7. INTERIM ANALYSES

Not applicable because, as this is a sponsor-open study, the sponsor will conduct unblinded reviews of the data during the course of the study for the purpose of safety assessment and facilitating dose-escalation decisions. In addition, these reviews may facilitate PK/PD modeling and/or supporting clinical development.

#### 8. REFERENCES

1. Pfizer Guidance for Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-antiarrhythmic Drugs; Members of the Cardiovascular Safety & Advisory Council (CVSAC); January 26, 2018.



# 9. APPENDICES



#### **Appendix 1. Summary of Efficacy Analyses**

Not Applicable fo this study

#### **Appendix 2. Data Derivation Details**

#### Appendix 2.1. Definition and Use of Visit Windows in Reporting

Not Applicable fo this study.

#### **Appendix 2.2. Endpoint Derivations**

Not Applicable fo this study

#### Appendix 2.3. Example SAS Code for Statistical Analyses

#### **Appendix 2.3.1. Analysis for DDI interaction (Part A):**

```
/* To compare Test PK Parameter to the Reference PK Parameter where l&var = log(&var)*

proc mixed data = input_dataset method = reml;
    class participant treatment period sequence;
    model l&var = treatment period sequence /ddfm = kr residual;
    random participant(sequence);
    lsmeans treatment;
    estimate 'trt1 - trt1' treatment -1 1 / cl alpha = 0.1;

run;
```

#### **Appendix 2.3.2. Analysis for DDI interaction (Part B):**

```
/* To compare Test PK Parameter to the Reference PK Parameter where l&var = log(&var)*
proc mixed data=tab.pk;
class Day Participant;
model l&var= Day / ddfm=KR;
random participant;
lsmeans Day;
Estimate 'Test vs Reference' Day -1 1 / cl alpha=0.1;
ods 'Estimates' out=est&var;
ods 'Ismeans' out=ls&var;
ods 'covparms' out=cov&var;
ods 'tests3' out=tst&var;
run;
```



# Appendix 3. List of Abbreviations

| Abbreviation | Term |
|---|---|
| Abs | absolute |
| AE | adverse event |
| ANCOVA | analysis of covariance |
| ANOVA | analysis of variance |
| aPTT | activated partial thromboplastin time |
| AUC | area under the plasma concentration-time curve |
| AUC <sub>12</sub> | area under the plasma concentration-time curve from time zero to |
| | time 12 hours post-dose |
| AUC <sub>24</sub> | area under the plasma concentration-time curve from time zero to |
| | time 24 hours post-dose |
| $AUC_{inf}$ | area under the plasma concentration-time curve from time zero |
| | extrapolated to infinite time |
| AUC <sub>last</sub> | area under the plasma concentration-time curve from time zero to the |
| | time of the last quantifiable concentration (C <sub>last</sub> ) |
| AV | atrioventricular |
| BLQ | below the limit of quantitation |
| BMI | body mass index |
| BP | blood pressure |
| bpm | beats per minute |
| CI | confidence interval |
| CK | creatine kinase |
| CKD-EPI | Chronic Kidney Disease Epidemiology Collaboration |
| CL/F | apparent oral clearance |
| $C_{max}$ | maximum plasma concentration |
| COVID-19 | coronavirus disease-19 |
| CP-I | Coproporphyrins I |
| CRF | case report form |
| CRO | contract research organization |
| CRU | clinical research unit |
| CSR | Clinical Study Report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CT | clinical trial |
| CV | coefficient of variation |
| DC | discontinuation |
| DDI | drug-drug interaction |
| DGAT | diacylglycerol acyltransferase |
| DILI | drug-induced liver injury |



| Abbreviation | Term |
|---|---|
| DMC | Data Monitoring Committee |
| DNA | deoxyribonucleic acid |
| EAC | event adjudication committee |
| EC | Ethics Committee |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| E-DMC | external data monitoring committee |
| EDP | exposure during pregnancy |
| EFD | embryo-fetal development |
| ET | early termination |
| EudraCT | European Clinical Trials Database |
| F/U | follow-up |
| FAP | final approved protocol |
| FAS | full analysis set |
| FDA | Food and Drug Administration |
| $f_{m}$ | fraction metabolized |
| FSBG | fingerstick blood glucose |
| FSH | follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transferase |
| GLIMMIX | generalized linear mixed-effects model with repeated measures |
| GLP | Good Laboratory Practice |
| GLP-1 | glucagon-like peptide 1 |
| GMC | geometric mean concentration |
| GMFR | geometric mean fold rise |
| GMR | geometric mean ratio |
| HAE | hypoglycemic adverse event |
| HbA1c | hemoglobin A1c |
| HDL-C | high density lipoprotein cholesterol |
| HR | heart rate |
| ICD | informed consent document |
| ICH | International Council for Harmonisation |
| IND | Investigational New Drug |
| INR | international normalized ratio |
| IP | investigational product |
| ITT | intent-to-treat |
| IV | intravenous(ly) |
| kel | elimination rate constant |
| Ki | apparent inactivation constant at half-maximal rate of inactivation |
| kinact | maximal inactivation rate |



| Abbreviation | Term |
|--------------|----------------------------------------------|
| LDL-C | low density lipoprotein cholesterol |
| LFT | liver function test |
| LLN | lower limit of normal |
| LLOQ | lower limit of quantitation |
| LOCF | last observation carried forward |
| LOD | limit of detection |
| LS | least-squares |
| LSM | least-squares mean |
| MAR | missing at random |
| MCH | mean corpuscular hemoglobin |
| MCHC | mean corpuscular hemoglobin concentration |
| MCV | mean corpuscular volume |
| MDR | multi-drug resistance |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MHP | mental health professional |
| mITT | modified intent-to-treat |
| MMRM | mixed-effects model with repeated measures |
| MMTT | mixed meal tolerance test |
| MNAR | missing not at random |
| CCI | |
| mRNA | messenger ribonucleic acid |
| msec | millisecond |
| MTD | maximum tolerated dose |
| N/A | not applicable |
| NAFLD | non-alcoholic fatty liver disease |
| NASH | non-alcoholic steatohepatitis |
| NNT | number needed to treat |
| NOAEL | no-observed-adverse-effect level |
| OAT | organic anion transporter |
| OATP | organic anion transporting polypeptide |
| OATP1B1 | organic anion transporting polypeptide 1B1 |
| OCT | organic cation transporter |
| PD | pharmacodynamic(s) |
| PHQ-9 | Patient Health Questionnaire-9 |
| PK | pharmacokinetic(s) |
| PLT | platelet |
| PP | per-protocol |
| PPAS | per-protocol analysis set |
| PR | pulse rate |
| PT | prothrombin time |



| Abbreviation | Term |
|---|---|
| PVC | premature ventricular contraction/complex |
| QT | time from beginning of the QRS complex to the end of the T wave |
| QTc | corrected QT |
| QTcF | corrected QT (Fridericia method) |
| qual | qualitative |
| Rac | accumulation ratio |
| RBC | red blood cells |
| RR | relative risk |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SGS | Statistical Guidance Standards |
| SoA | Schedule of Activities |
| SOP | standard operating procedure |
| SRSD | single reference safety document |
| SToD | study team on demand |
| SUSAR | suspected unexpected serious adverse reaction |
| t <sub>1/2</sub> | terminal half-life |
| T4 | thyroxine |
| TA | therapeutic area |
| TBA | total bile acids |
| TEAE | treatment-emergent adverse event |
| TG | triglycerides |
| THC | tetrahydrocannabinol |
| $T_{\text{max}}$ | time for C <sub>max</sub> |
| TSH | thyroid-stimulating hormone |
| ULN | upper limit of normal |
| US | United States |
| V <sub>z</sub> /F | apparent oral volume of distribution |
| WBC | white blood cell |
| WHO | World Health Organization |
| WHODD | World Health Organization Drug Dictionary |
| WOCBP | woman of childbearing potential |



# Appendix 4. Categorical Classes for ECG and Vital Signs of Potential Clinical Concern

## **Categories for QTcF**

| Absolute value of QTcF (msec) | >450 and ≤480 | >480 and ≤500 | >500 |
|--------------------------------|---------------|---------------|------|
| Increase from baseline in QTcF | >30 and ≤60 | >60 | |
| (msec) | | | |

### Categories for PR and QRS

| PR (ms) | max. ≥300 | |
|------------------|---------------|-------------------|
| PR (ms) increase | Baseline >200 | Baseline ≤200 and |
| from baseline | and max. | max. ≥50% |
| | ≥25% increase | increase |
| QRS (ms) | max. ≥140 | |
| QRS (ms) | ≥50% increase | |
| increase from | | |
| baseline | | |

### **Categories for Vital Signs**

| Systolic BP (mm Hg) | min. <90 | |
|---------------------------|-------------------|-------------------|
| Systolic BP (mm Hg) | max. decrease ≥30 | max. increase ≥30 |
| change from baseline | | |
| Diastolic BP (mm Hg) | min. <50 | |
| Diastolic BP (mm Hg) | max. decrease ≥20 | max. increase ≥20 |
| change from baseline | | |
| Supine pulse rate (bpm) | min. <40 | max. >120 |
| Standing pulse rate (bpm) | min. <40 | max. >140 |



# Appendix 5. C-SSRS Mapped to C-CASA - Suicidal Ideation and Behavior Events and Codes

Table 1. C-SSRS Mapped to C-CASA (Suicidality Events and Codes)

| Event | | |
|---|---|---|
| Code | | C-SSRS Response |
| Suicid | Suicidal Ideation | |
| 1 | Passive | "Yes" on "Wish to be dead" |
| 2 | Active: Nonspecific (no method, intent, or plan) | "Yes" on "Non-Specific Active Suicidal |
| | | Thoughts" |
| 3 | Active: Method, but no intent or plan | "Yes" on "Active Suicidal Ideation with |
| | | Any Methods (Not Plan) without Intent to |
| | | Act" |
| 4 | Active: Method and intent, but no plan | "Yes" on "Active Suicidal Ideation with |
| | | Some Intent to Act, without Specific Plan" |
| 5 | Active: Method, intent, and plan* | "Yes" on "Active Suicidal Ideation with |
| | | Specific Plan and Intent" |
| Suicidal Behavior | | |
| 1 | Completed suicide | "Yes" on "Completed Suicide" |
| 2 | Suicide attempt | "Yes" on "Actual Attempt" |
| 3 | Interrupted attempt | "Yes" on "Interrupted attempt" |
| 4 | Aborted attempt | "Yes" on "Aborted attempt" |
| 5 | Preparatory actions toward imminent suicidal | "Yes" on "Preparatory Acts or Behavior" |
| | behaviors | |
| Self-injurious behavior, no suicidal intent | | |
| | Self-injurious behavior, no suicidal intent | "Yes" on "Has subject engaged in Non- |
| | | suicidal Self-Injurious Behavior?" |

\*According to C-SSRS, the definition of *plan* includes intent (i.e., intent to complete the suicide is implicit with the concept of plan). Thus, there is no need for the category *method and plan, but no intent*